CLINICAL TRIAL: NCT00083863
Title: Framingham: Inflammation, Genes & Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Emelia Benjamin, Principle Investigator, Boston University
Other Study IDs: 1257; R01HL076784 (NIH)
Record Dates: First submitted 2004-06-02; First posted 2004-06-04 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Inflammation
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (2):
- Framingham Heart Study Offspring
- FHS Gen 3

SUMMARY:
To investigate the contribution of genetic and environmental factors to vascular inflammation, and to define the extent to which inflammatory phenotypes and genotypes predict subclinical and clinical cardiovascular disease (CVD).

DETAILED DESCRIPTION:
BACKGROUND:

Recent experimental and clinical studies support the concept that vascular inflammation is central to the development of atherosclerosis, and that systemic inflammatory markers predict a wide array of cardiovascular disease (CVD) events. There is increasing interest in the role of genetic variation in inflammation contributing to the susceptibility for CVD. To date mostly small case-control studies have suggested that polymorphisms in inflammatory genes are associated with subclinical and clinical CVD, but the studies have differed with regard to which genes are central. The investigators have previously measured systemic markers of vascular inflammation (e.g. CRP, sICAM-1, MCP-1, IL-6) and oxidative stress (isoprostanes), in a population-based sample of 3800 middle-aged and elderly men and women of the Framingham Heart Study offspring cohort. They now propose to genotype inflammatory candidate genes in the Framingham offspring cohort which have been phenotyped for CVD risk factors, subclinical CVD.They also propose to measure systemic inflammatory markers in the Framingham Study Generation III cohort, who are the children of the offspring cohort.

DESIGN NARRATIVE:

Dr. Benjamin and colleagues will genotype inflammatory candidate genes in the Framingham offspring cohort which have been phenotyped for CVD risk factors, subclinical CVD. They also will measure systemic inflammatory markers in the Framingham Study Generation III cohort, who are the children of the offspring cohort. The central hypothesis of this study is that systemic vascular inflammation represents a complex phenotype that evolves over a lifetime and is influenced by both environmental and genetic factors. They further postulate that variations in the inflammatory phenotype (marker levels) and genotype predispose to the development of CVD. The purpose of this study is to determine the contribution of genetic and environmental factors to vascular inflammation, and to define the extent to which inflammatory phenotypes and genotypes predict subclinical and clinical CVD, and enhance risk prediction models. The specific aims are: Aim 1. To examine the environmental determinants of systemic inflammation in the community. Aim 2. To investigate the genetic determinants of systemic inflammation. Aim 3. To identify the inflammatory phenotypic and genetic determinants of subclinical CVD. Aim 4. To determine the contribution of inflammatory phenotype versus genotype to prevalent and incident CVD and to incident hypertension. The investigation will increase understanding as to whether inflammation is a core risk factor for CVD or is merely a marker of presence and burden of other CVD risk factors. These insights will fundamentally contribute to knowledge about the pathophysiology of CVD and may lead to improved prevention, risk stratification and management of CVD.

ELIGIBILITY:
Offspring & Generation 3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Observational Cohort Study
Sampling Method: Non-Probability Sample
Enrollment: 7374 (Actual)
Dates: Start 2004-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Cardiovascular diseases | The FHS study is longitudinal so events will accrue over decades of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Emelia Benjamin, Principal Investigator — Boston University